CLINICAL TRIAL: NCT05523284
Title: Transvaginal Ultrasound-guided Culdocentesis for Peritoneal Fluid Cytokines in Patients With Possible Superficial Endometriosis But no Ultrasound-diagnosed Ovarian or Deep Endometriosis (SPG)
Brief Title: Combining Ultrasound and Biomarkers to Diagnose Superficial Endometriosis
Acronym: SPGENDO
Status: Enrolling by invitation | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: LRG - SPGENDO
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis (Diagnosis); Endometriosis
Keywords: Endometriosis; Diagnosis; Ultrasound; Biomarkers
MeSH Terms: conditions — Endometriosis; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — SPG fluid (flushed saline) will be aspirated from the POD and evaluated using full proteomic and genomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SonoPODography — SonoPODography (SPG) is a novel ultrasound-guided technique whereby saline is injected through the cervix and flushed into the POD, creating an acoustic window for diagnosing superficial endometriosis.

SUMMARY:
Endometriosis is a benign gynecological disease characterized by uterine-like cells growing outside the uterus, leading to pain, infertility, and inflammation. Endometriosis most commonly occurs in the forms of Superficial Endometriosis (SE), Deep Endometriosis and Ovarian Endometriosis (Endometrioma) (OE). Ultrasound diagnosis of DE and OE has become more reliable with advances in ultrasound technology, technique and expertise, leading to decreased diagnosis time for patients and allowing for better optimization of surgeries if required. SE, however, lacks any reliable non-invasive diagnosis methods.

SE is the most common form of endometriosis and is defined as a disease that lines the peritoneum and is small and superficial in nature, leading to chronic inflammation, infertility, and pain. SE is difficult to visualize on ultrasound due to its size and alignment with tissue, requiring fluid to expand the pelvis and partially suspend these small lesions, allowing them to be diagnosed through ultrasound. Leonardi et al. observed that in some patients, a physiologic change occurs whereby fluid fills the pouch of Douglas (POD), allowing increased visualizing during ultrasound. This led to the development of Saline-infused sonoPODgraphy (SPG), a novel method utilizing modified commonly used ultrasound techniques called saline-infusion sonohysterography (SIS) and hysterosalpingo-contrast-sonography (HyCoSy), to reliably visualize the POD (Leonardi et al, 2019). Visualizing the POD is important as SE is often deposited in the POD.

This diagnostic accuracy pilot study aims to pioneer the technique whereby SPG will be evaluated as a novel, rapid, non-invasive diagnostic tool for SE. The injected fluid from the POD will be withdrawn and evaluated for novel biomarkers, allowing us to further develop rapid diagnostics and better understand disease mechanisms. We hypothesize that SPG will allow for the diagnosis of SE with a diagnostic accuracy parallel to the current invasive gold standard, laparoscopy.

DETAILED DESCRIPTION:
Introduction Endometriosis is a common benign disease characterized by the growth of uterine cells outside of the uterus, causing various forms of pelvic pain and/or difficulty with conceiving a pregnancy, amongst other symptoms. Endometriosis most commonly occurs in the forms of Superficial Endometriosis (SE), Deep Endometriosis and Ovarian Endometriosis (Endometrioma) (OE). Ultrasound diagnosis of DE and OE has become more reliable with advances in ultrasound technology, technique and expertise leading to decreased diagnosis time for patients and allowing for better optimization of surgeries if required. SE, however, lacks any reliable non-invasive diagnosis methods.

SE is the most common form of endometriosis and is defined as a disease that lines the peritoneum and is small and superficial in nature, leading to chronic inflammation, infertility, and pain. SE is difficult to visualize on ultrasound due to its size and alignment with tissue, requiring fluid in order expand the pelvis and partially suspend these small lesions, allowing them to be diagnosed through ultrasound. Leonardi et al. observed that in some patients, a physiologic change occurs whereby fluid fills the pouch of Douglas (POD) allowing increased visualizing during ultrasound. This led to the development of Saline-infused sonoPODgraphy (SPG), a novel method utilizing modified commonly used ultrasound techniques called saline-infusion sonohysterography (SIS) and hysterosalpingo-contrast-sonography (HyCoSy), to reliably visualize the POD. The ability to visualize the POD is important as SE is often deposited in the POD.

Biomarkers are also an active area of research in endometriosis diagnosis. There are possible biomarkers that have been identified in the peritoneal fluid of people with endometriosis, including Tumour Necrosis Factor (TNF) and interleukin-6 (IL-6). Indeed, a landmark biomarker study in 2002 demonstrated that TNF in peritoneal fluid had a 100% sensitivity for identifying women with endometriosis. However, this finding has never been further evaluated or validated, even though there is evidence of TNF involvement in endometriosis development. Recently, insulin-like growth factor 1 (IGF-1) has been noted to be elevated in the peritoneal fluid of people with endometriosis compared to those without. Further, IGF-1 has also been found to contribute to the development of abnormal nerves, which may explain the link between endometriosis and pain.

The previous work with POD imaging combined with the knowledge of endometriosis biomarkers leads to the question: Can these non-invasive diagnostic methods be combined to diagnose superficial endometriosis accurately and consistently. We hypothesize that using a combined approach of SPG and biomarker analysis to diagnose superficial endometriosis will provide sufficient evidence to support a large multi-centre international diagnostic accuracy trial.

Technical Study Summary

Study Design

This diagnostic accuracy feasibility study is a Health Canada-sponsored study whereby fluid will be injected through the cervix among recruited and consented participants. During routine clinical visits at the McMaster Women's Health Clinic, participants will be recruited on a rolling basis. The study will start in October 2022 and will continue until the intended sample size is reached and/or January 2024

Sample size

In this feasibility trial, we aim to recruit all patients who meet the eligibility criteria over 14 months from the McMaster University Medical Center. Given the previous publication on SPG and SE by Leonardi et al (2020), based on an estimated prevalence of SE of 60 % and sensitivity of 80 %, and a half-width of 95 % CI of 0.15 (i.e. the sensitivity cannot be lower than 0.65), a total of 50 participants will be required.

Variables

In addition to data regarding index and reference standard tests, demographic and clinical information that is routinely collected will be obtained, including age, BMI, gravidity, parity, history of infertility (as defined by 1 year of trying to conceive without success), past medical history, past surgical history, use of hormonal agents for contraception or treatment of gynecological concern, menstrual characteristics (last menstrual period (at time of TVS-C and surgery), cycle frequency, duration of menses, abnormal uterine bleeding). Previous sexually transmitted and blood-borne infections (STBBI) results will be assessed as potential differential diagnoses when adhesions are present in the absence of endometriosis upon surgery.

During TVS, the disease will be characterized for each patient using the Leonardi et al (2020) modified descriptors for SE under TVS, including size, location, hyperechoic projections, hypoechoic areas, cystic areas, filmy adhesions, peritoneal pockets, and jiggling of the lesion. These characteristics will then be compared to surgical findings using the validated and internationally recognized WERF Surgical questionnaire as categorical data. Due to previous findings in the Leonardi et al (2020) study suggests that SPG may be unsuccessful (SPG fluid filling the POD) in a small portion of the population (5.6%; excluding those with POD obliteration), and the rate of success will be recorded and reported as part of the diagnostic accuracy and indicative of the efficacy of the technique. However, in the event of unsuccessful SPG, tubal patency assessment will be performed at laparoscopy with dye chromotubation to assess whether the bilateral tubal blockage was the reason for the failure of SPG. As there is a slight possibility of having physiological fluid accumulated in the POD before SPG, an estimate of volume will be made under TVS for those with fluid present (calculated using a length x width x height approach, which is the generally accepted method to calculate the volume of pelvic fluid). The volume of SPG fluid injected will be recorded as a continuous variable for each participant. Upon the completion of the study, the volumes will be categorized into groups, allowing for subgroup analysis.

Following the TVS-C, participants will be asked to complete a short questionnaire on their tolerability and acceptance of the procedure. Similarly, following laparoscopy, patients will be asked to answer the same series of questions regarding the laparoscopy and to re-evaluate the TVS-C, having had both procedures to compare.

Statistical analysis

Sensitivity, specificity, positive, and negative predictive values will be calculated for SPG and identified biomarkers in the aspirated fluid. The demographic and clinical variables, peritoneal fluid features and TNF levels, TVS and surgical findings will be described descriptively using standardized terminology for all participants per routine clinical guidelines and assessed as categorical data upon data cleaning. The success of the acquisition of peritoneal fluid will be described. Subgroup analysis will be done with those who had serosanguinous peritoneal fluid.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years of Age
* Assigned Female at Birth
* Confirmed or Suspected Case of Superficial Endometriosis
* Willing and Able to Provide Informed Written Consent

Exclusion Criteria:

* Pre-Menarche or Post-Menopausal
* No History of Vaginal Penetration / Intercourse
* Concern for pre-malignancy or presence/history of malignancy
* Known Bleeding Disorder
* Presence of Deep or Ovarian Endometriosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited from the McMaster Women's Health Clinic during routine pelvic evaluation using transvaginal ultrasound to assess the pelvic and abdominal cavity for any pathologies. Only participants with a uterus (assigned female at birth) will be eligible to join the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Determine the diagnostic accuracy of SPG as a non-invasive diagnostic modality for superficial endometriosis, in the absence of DE, OE, and POD obliteration. | 2022-2024
  The diagnostic accuracy of SPG and biomarkers will be compared to the current gold standard, laparoscopy and histology.

SECONDARY OUTCOMES:
1. Characterize superficial endometriosis under TVS using modified descriptors from the Leonardi et al (2020) SPG study. | 2022-2024
  Superficial endometriosis will be characterized and described using the developed standardised terminology by Leonardi et al (2020), to assist in the development of an international consensus.
2. Determine the association between TVS and surgical characteristics of superficial endometriosis using the accepted World Endometriosis Research Foundation (WERF) guidelines | 2022-2024
  The characterization of superficial endometriosis during laparoscopy will be conducted using the WERF guidelines and compared to the descriptors used during ultrasound.
3. Assess the tolerability and acceptance of SPG as a rapid, non-invasive diagnostic technique for SE among those with endometriosis using a questionnaire | 2022-2024
  A questionnaire will be used to evaluate the tolerability to efficacy of SPG using a 10-point Likert Scale (1 = almost no pain, 10 = worst pain ever experienced in life)
4. Externally validate the Determine the rate of success rate of SPG (fluid filling the POD) from a technicity perspective | 2022-2024
  The success rate will be determine by the ability of SPG fluid to enter and fill the POD, further illustrating the efficacy of the technique.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Leonardi M, Robledo KP, Espada M, Vanza K, Condous G. SonoPODography: A new diagnostic technique for visualizing superficial endometriosis. Eur J Obstet Gynecol Reprod Biol. 2020 Nov;254:124-131. doi: 10.1016/j.ejogrb.2020.08.051. Epub 2020 Sep 16. PMID 32961428
- [Result] Chapron C, Tosti C, Marcellin L, Bourdon M, Lafay-Pillet MC, Millischer AE, Streuli I, Borghese B, Petraglia F, Santulli P. Relationship between the magnetic resonance imaging appearance of adenomyosis and endometriosis phenotypes. Hum Reprod. 2017 Jul 1;32(7):1393-1401. doi: 10.1093/humrep/dex088. PMID 28510724
- [Result] Cheong YC, Shelton JB, Laird SM, Richmond M, Kudesia G, Li TC, Ledger WL. IL-1, IL-6 and TNF-alpha concentrations in the peritoneal fluid of women with pelvic adhesions. Hum Reprod. 2002 Jan;17(1):69-75. doi: 10.1093/humrep/17.1.69. PMID 11756364
- [Result] Deslandes A, Parange N, Childs JT, Osborne B, Bezak E. Current Status of Transvaginal Ultrasound Accuracy in the Diagnosis of Deep Infiltrating Endometriosis Before Surgery: A Systematic Review of the Literature. J Ultrasound Med. 2020 Aug;39(8):1477-1490. doi: 10.1002/jum.15246. Epub 2020 Feb 21. PMID 32083336
- [Result] Forster R, Sarginson A, Velichkova A, Hogg C, Dorning A, Horne AW, Saunders PTK, Greaves E. Macrophage-derived insulin-like growth factor-1 is a key neurotrophic and nerve-sensitizing factor in pain associated with endometriosis. FASEB J. 2019 Oct;33(10):11210-11222. doi: 10.1096/fj.201900797R. Epub 2019 Jul 10. PMID 31291762
- [Result] Goncalves MO, Siufi Neto J, Andres MP, Siufi D, de Mattos LA, Abrao MS. Systematic evaluation of endometriosis by transvaginal ultrasound can accurately replace diagnostic laparoscopy, mainly for deep and ovarian endometriosis. Hum Reprod. 2021 May 17;36(6):1492-1500. doi: 10.1093/humrep/deab085. PMID 33864088
- [Result] Leonardi M, Espada M, Lu C, Stamatopoulos N, Condous G. A Novel Ultrasound Technique Called Saline Infusion SonoPODography to Visualize and Understand the Pouch of Douglas and Posterior Compartment Contents: A Feasibility Study. J Ultrasound Med. 2019 Dec;38(12):3301-3309. doi: 10.1002/jum.15022. Epub 2019 May 15. PMID 31090229
- [Result] Piessens S, Edwards A. Sonographic Evaluation for Endometriosis in Routine Pelvic Ultrasound. J Minim Invasive Gynecol. 2020 Feb;27(2):265-266. doi: 10.1016/j.jmig.2019.08.027. Epub 2019 Sep 4. PMID 31493569
- [Result] Reis FM, Santulli P, Marcellin L, Borghese B, Lafay-Pillet MC, Chapron C. Superficial Peritoneal Endometriosis: Clinical Characteristics of 203 Confirmed Cases and 1292 Endometriosis-Free Controls. Reprod Sci. 2020 Jan;27(1):309-315. doi: 10.1007/s43032-019-00028-1. Epub 2020 Jan 1. PMID 32046376
- [Result] Vercellini P, Vigano P, Somigliana E, Fedele L. Endometriosis: pathogenesis and treatment. Nat Rev Endocrinol. 2014 May;10(5):261-75. doi: 10.1038/nrendo.2013.255. Epub 2013 Dec 24. PMID 24366116
- [Result] Vitonis AF, Vincent K, Rahmioglu N, Fassbender A, Buck Louis GM, Hummelshoj L, Giudice LC, Stratton P, Adamson GD, Becker CM, Zondervan KT, Missmer SA; WERF EPHect Working Group. World Endometriosis Research Foundation Endometriosis Phenome and Biobanking Harmonization Project: II. Clinical and covariate phenotype data collection in endometriosis research. Fertil Steril. 2014 Nov;102(5):1223-32. doi: 10.1016/j.fertnstert.2014.07.1244. Epub 2014 Sep 22. PMID 25256930
- [Result] Zondervan KT, Becker CM, Missmer SA. Endometriosis. N Engl J Med. 2020 Mar 26;382(13):1244-1256. doi: 10.1056/NEJMra1810764. No abstract available. PMID 32212520